CLINICAL TRIAL: NCT03913923
Title: International Multicenter Double-Blind Placebo-Controlled Comparative Randomized Trial of Efficacy and Safety of BCD-217 (Anti-CTLA-4 and Anti-PD-1) And BCD-100 (Anti-PD-1) Therapy Compared to BCD-100 Monotherapy as First-Line Treatment in Patients With Unresectable or Metastatic Melanoma
Brief Title: Study of Efficacy and Safety of BCD-217 (Anti-CTLA-4 and Anti-PD-1) Followed By BCD-100 (Anti-PD-1) Versus BCD-100 Monotherapy as First-Line Treatment in Patients With Unresectable or Metastatic Melanoma
Acronym: OBERTON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-217-1
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Melanoma; Melanoma Metastatic
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-217 and BCD-100 (Experimental): Patients will receive 4 blinded infusions of BCD-217 plus Placebo. Starting with the fith infusion patients will receive unblinded BCD-100 monotherapy.
  Interventions: Biological: BCD-217; Biological: BCD-100; Other: Placebo
- BCD-100 monotherapy (Active Comparator): Patients will receive 4 blinded infusions of BCD-100 plus Placebo. Starting with the fith infusion patients will receive unblinded BCD-100 monotherapy.
  Interventions: Biological: BCD-100; Other: Placebo

INTERVENTIONS:
Biological: BCD-217 — Combination of anti-CTLA-4 and anti-PD-1 monoclonal antibodies, 1mg/kg and 3 mg/mg, respectively, given Q3W as IV infusion for first 4 blinded infusions
  Arms: BCD-217 and BCD-100
Biological: BCD-100 — Anti-PD-1 monoclonal antibody, 3 mg/kg, given Q3W as IV infusion for first 4 blinded infusions, after - 1 mg/kg, given Q2W as IV infusion
Other: Placebo — Placebo

SUMMARY:
This is a multicenter randomized double-blind placebo-controlled phase II clinical trial. The purpose of this trial is to evaluate efficacy and safety of therapy consisting of BCD-217 (fixed dose combination of anti-CTLA-4 and anti-PD-1 monoclonal antibodies) and sequential BCD-100 (anti-PD-1 monoclonal antibody) versus BCD-100 monotherapy as first-line treatment in patients with treatment-naïve unresectable or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form and the subject's ability to follow the Protocol requirements;
2. Age: 18 years and older at the signing of the informed consent;
3. Histologically verified (documented) melanoma;
4. Previously untreated unresectable stage III melanoma or metastatic stage IV melanoma;
5. Available tissue blocks for histological examination or patient's agreement to give biopsy specimens
6. Patient's consent for PD-L1 expression status and BRAF V600 testing;
7. ECOG performance status of 0 or 1;
8. Life expectancy of at least 12 weeks from the screening;
9. At least one RECIST 1.1-defined measurable target lesion confirmed by an independent review;
10. Patients with reproductive potential must agree to practice acceptable methods of birth control throughout the entire trial period, starting from signing the informed consent and up to 24 weeks after the last dose of investigational drug.

Exclusion Criteria:

1. Indications for radical (surgical, radiation) therapy;
2. A history of previous systemic antitumor therapy for unresectable or metastatic melanoma ;
3. Prior therapy with checkpoint inhibitors (e.g., anti-CTLA-4 and/or anti-PD-1/PD-L1/PD-L2 products);
4. Prior therapy with BRAF and MEK protein kinase inhibitors;
5. Use of immunostimulants, monoclonal antibodies and/or colony-stimulating factors within less than 4 weeks prior to randomization in the study;
6. Ocular melanoma;
7. Mucosal melanoma;
8. CNS metastases;
9. Impossibility to determine PD-L1 status and/or BRAF status;
10. Subjects with severe comorbidities, life-threatening acute complications of the primary disease (including massive pleural, pericardial, or peritoneal effusions requiring intervention , pulmonary lymphangitis, bleeding, or organ perforation) at the time of signing the informed consent form;
11. Ongoing concomitant diseases at the time of screening, which increase the risk of severe adverse events during the administration of the study therapy:

    * stable angina, functional class III-IV,
    * unstable angina or a history of myocardial infarction within less than 6 months prior to signing the informed consent form;
    * moderate to severe heart failure (classes III and IV according to NYHA classification);
    * uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg) ;
    * a history of atopic asthma , angioedema;
    * respiratory failure (moderate to severe), grade 3 or 4 chronic obstructive pulmonary disease;
    * any other concomitant diseases (including, but not limited to, metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, gastrointestinal disorders), which expose the patient to an unacceptable risk during the study therapy;
12. Known or suspected systemic autoimmune diseases (including, but not limited to, systemic lupus erythematosus, Crohn's disease, nonspecific ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.) ;
13. History of interstitial pulmonary disease or pneumonitis requiring systemic glucocorticoids;
14. The need for glucocorticoid therapy (at >10 mg/day prednisolone equivalent doses) or any other drugs with immunosuppressive effects within 14 days prior to randomization;
15. Hematologic abnormalities :

    * neutrophils <1.5×109/L,
    * platelets <100×109/L,
    * hemoglobin <90 g/L;
16. Renal impairment: creatinine ≥2.5×ULN;
17. Hepatic impairment :

    * total bilirubin ≥3×ULN (except for the patients with Gilbert's syndrome, in whom bilirubin levels should not exceed 50 μmol/L),
    * AP, AST or ALT ≥2.5×ULN (≥5×ULN in case of patients with liver metastases);
18. Any antitumor treatment within less than 4 weeks or surgery within less than 28 days prior to randomization within the study;
19. History of oncological disease, except for radically treated diseases with remission for over 5 years prior randomization in this study ;
20. Conditions limiting the patient's ability to comply with the Protocol requirements (in the Investigator's opinion );
21. Participation in other clinical studies within less than 30 days prior to randomization and during this clinical study ;
22. Acute infections or activation of chronic infectious diseases or systemic antibacterial therapy within less than 28 days prior to randomization;
23. Active hepatitis B, active hepatitis C (confirmed by PCR), active syphilis, HIV-infection, currently or previously ;
24. Impossibility to administer the investigational product intravenously;
25. Impossibility to administer intravenous contrast agents (including due to hypersensitivity to contrast media);
26. Hypersensitivity to any of the components of BCD-100 or BCD-217;
27. A history of hypersensitivity to monoclonal antibody products;
28. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival | 2 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  The time from the date of randomization until progression of disease per RECIST 1.1 and iRECIST or death
Overall Survival (OS) | 2 years
  The time from the date of randomization until death
Overall Response Rate | 2 years
  The percentage of the participants who have a Complete Response or a Partial Response as assessed by a blind independent central reviewer per RECIST 1.1. and iRECIST
Disease Control Rate | 2 years
  The percentage of the participants who have a Complete Response, a Partial Response or a Stable DIsease as assessed by a blind independent central reviewer per RECIST 1.1. and iRECIST
Time to Response (TTR) | 2 years
  TTR will be calculated from the randomization date
Duration of Response | 2 years
  DOR will be calculated from the moment of registration of response till event (progression or death)

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (23):
- Belarus (2):
  - State Institution "N.N. Aleksandrov Republican Research and Practical Center for Oncology and Medical Radiology", The Settlement of Lesnoy, Minsk District
  - Healthcare Institution "Minsk Municipal Clinical Oncolo-gy Dispensary" (MMCOD), Minsk
- Russia (21):
  - Clinical Oncologic Dispensary No. 2, Sochi, Krasnodar Territory
  - Krasnoyarsk Regional Clinical Oncological Dispensary named after A.I. Kryzhanovsky, Krasnoyarsk, Krasnoyarsk Krai
  - Murmansk Regional Clinical Hospital named after P.A. Bayandina, Murmansk, Murmansk Oblast
  - LLC "New Clinic", Pyatigorsk, Stavropol Kray
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - State Budgetary Healthcare Institution of the Ar-khangelsk Region "Arkhangelsk Clinical Oncology Dispensary", Arkhangelsk
  - Territorial State Budgetary Healthcare Institution "Altai Territorial Clinical Oncology Dispensary", Barnaul
  - State Budgetary Healthcare Institution "Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine",, Chelyabinsk
  - State public health institution "Republican Clinical Oncology Dispensary" of the Ministry of Health of the Republic of Tatarstan, Kazan'
  - Regional State Budgetary of Healthcare Insti-tution "Kostroma Oncology Dispensary", Kostroma
  - Medsi Group of Companies Joint-Stock Company, Moscow
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - State Health Care Institution "Moscow City Oncology Hospital № 62" Moscow Health Department, Moscow
  - State Budgetary Healthcare Institution of the Novosi-birsk Region "Novosibirsk Regional Clinical Oncolo-gy Dispensary", Novosibirsk
  - State budget healthcare institution Omsk region "Clinical Oncology Dispensary", Omsk
  - JSC "Modern Medical Technologies", Saint Petersburg
  - AV Medical Group Limited Liability Company, Saint Petersburg
  - Federal State Institution "N.N. Petrov National Medical Research Center for Oncology", Saint Petersburg
  - Saint-Petersburg Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "St. Petersburg State University", Saint Petersburg
  - State-financed Health Institution "Samara Region Clinical Oncology Dispansary", Samara

IPD SHARING:
Plan to Share IPD: No